CLINICAL TRIAL: NCT00055653
Title: Unrelated Umbilical Cord Blood As An Alternate Source Of Stem Cells Transplantation
Brief Title: Donor Umbilical Cord Blood Transplantation in Treating Patients With Leukemia, Lymphoma, or Nonmalignant Hematologic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Philip McCarthy, Roswell Park Cancer Institute
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270487; RPCI-DS-00-22
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases
Keywords: refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; chronic myelomonocytic leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; acute undifferentiated leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Biphenotypic, Acute; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Antilymphocyte Serum; Filgrastim; Busulfan; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Melphalan; Methylprednisolone; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: melphalan
Drug: methylprednisolone
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Umbilical cord blood transplantation may be able to replace immune cells that were destroyed by the chemotherapy or radiation therapy that was used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of allogeneic umbilical cord blood transplantation in treating patients who have leukemia, lymphoma, or nonmalignant hematologic disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine 180-day survival in patients with malignant or nonmalignant hematologic diseases treated with allogeneic umbilical cord blood transplantation. (Severe aplastic anemia, Fanconi anemia, and marrow failure syndromes strata are closed to accrual; adult [over 18 years of age] patient stratum is closed to accrual.)
* Determine disease-free and long-term survival in patients treated with this regimen.
* Determine the incidence of neutrophil engraftment, primary and secondary graft failure, platelet engraftment, and red blood cell engraftment in patients treated with this regimen.
* Determine the incidence and severity of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine the incidence of complications, including infection, veno-occlusive disease, and interstitial pneumonitis, in patients treated with this regimen.
* Determine the incidence of relapse, other malignancies, lymphoproliferative disorders, and posttransplantation myelodysplasia in patients treated with this regimen.
* Determine the immune reconstitution in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are grouped according to the following strata:

* Stratum I: Malignant disease, 5/6 or 6/6 HLA match, age 18 and under
* Stratum II: Malignant disease, 4/6 HLA match, age 18 and under
* Stratum III: Malignant disease, 3/6 HLA match, age 18 and under
* Stratum IV: Malignant disease, 2/6 or 1/6 HLA match, age 18 and under
* Stratum V (closed to accrual): Severe aplastic anemia, Fanconi anemia, or other marrow failure syndrome
* Stratum VI: Inborn errors of metabolism/storage diseases and other nonmalignant diseases not included in stratum V
* Stratum VII: Malignant disease receiving alternative conditioning regimen comprising busulfan and melphalan
* Stratum VIII (closed to accrual): Adult patients (over age 18)
* Conditioning therapy: Patients are assigned to 1 of 5 groups according to diagnosis.

  * Group I (malignant disease or severe aplastic anemia [severe aplastic anemia closed to accrual]): Patients undergo total body irradiation (TBI) once or twice daily on days -8 to -4. Patients then receive cyclophosphamide IV on days -3 and -2, methylprednisolone IV on days -3 to 0, and antithymocyte globulin (ATG) IV once or twice daily on days -3 to -1.
  * Group II (Fanconi anemia [closed to accrual]): Patients undergo TBI on day -6, and then receive cyclophosphamide IV and fludarabine IV on days -5 to -2, and methylprednisolone IV and ATG IV on days -5 to -1.
  * Group III (inborn errors of metabolism/storage disease): Patients receive oral busulfan 4 times daily on days -9 to -6, cyclophosphamide as in group II, and methylprednisolone and ATG as in group I.
  * Group IV (other nonmalignant diseases): Patients receive conditioning therapy as in group III. Patients with familial erythrophagocytic lymphohistiocytosis or Langerhans cell histiocytosis also receive etoposide on days -5 to -3.
  * Group V (non-TBI regimen for leukemia patients under 2 years of age): Patients receive oral busulfan 4 times daily on days -8 to -5, melphalan IV on days -4 to -2, and methylprednisolone and ATG as in group I.
* Allogeneic umbilical cord blood transplantation: All patients undergo umbilical cord blood transplantation on day 0. Beginning on day 0 or 1, patients receive filgrastim (G-CSF) IV or subcutaneously daily until blood counts recover.
* Graft-versus-host disease prophylaxis: Patients receive cyclosporine (IV or oral) beginning between days -3 and -1 and continuing for 1 year after transplantation and methylprednisolone twice daily beginning on day 1 and continuing until blood counts recover.

Patients are followed weekly for 14 weeks, at 100 days, and at 4, 5, 6, 9, 12, 18, 24, and 36 months.

PROJECTED ACCRUAL: A total of 360 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia (AML)*

    * With or without history of myelodysplastic syndromes (MDS)
    * Patients in first complete remission (CR) (no greater than 5% blasts in marrow) with translocations t(8;21) and inv(16) are allowed provided they failed first-line induction therapy
    * Patients in first CR (no greater than 5% blasts in marrow) with translocations t(15;17) are allowed provided at least 1 of the following is true:

      * Failed first-line induction therapy
      * Molecular evidence of persistent disease
    * No patients in first CR and with Down syndrome
  * Acute lymphoblastic leukemia (ALL)*, meeting 1 of the following criteria:

    * Not in first CR (no greater than 5% blasts in marrow)
    * In first CR and high risk as defined by 1 of the following:

      * Hypoploidy (no more than 44 chromosomes)
      * Pseudodiploidy with translocations or molecular evidence of t(9;22), 11q23, or t(8;14) (excluding B-ALL) or +MLL gene rearrangement
      * One of the following elevated WBC levels:

        * WBC greater than 100,000/mm^3 if 6 to 12 months of age
        * WBC greater than 200,000/mm^3 if between 10 and 17 years of age
        * WBC greater than 20,000/mm^3 if 18 years of age and over (adult [over 18 years of age] patient stratum closed to accrual)
      * Failed to achieve CR after 4 weeks of induction therapy
    * B-ALL that is not in first CR or that meets at least 1 of the high-risk criteria specified above

      * No translocation t(8;14)
      * No blasts with surface immunoglobulins
      * CD10 negative
  * Undifferentiated leukemia*
  * Infant leukemia*
  * Biphenotypic leukemia*
  * Chronic myelogenous leukemia, meeting 1 of the following criteria:

    * Accelerated phase
    * Chronic phase

      * At least 1 year from diagnosis without an identified matched unrelated bone marrow donor AND unresponsive to or unable to tolerate interferon
    * Blast crisis* (greater than 30% promyelocytes plus blasts in the marrow)
  * One of the following MDS:

    * Refractory anemia
    * Refractory anemia with ringed sideroblasts
    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
  * Paroxysmal nocturnal hemoglobinuria
  * Hodgkin's or non-Hodgkin's lymphoma beyond first CR or failed primary induction therapy

    * Tumor displays chemosensitivity (greater than 50% reduction in mass size after the most recent therapy) NOTE: *Patients in third or greater medullary relapse or refractory disease (other than primary induction failures) or blast crisis receive the study busulfan/melphalan conditioning regimen)

OR

* Diagnosis of one of the following nonmalignant diseases :

  * Acquired severe aplastic anemia (stratum closed to accrual)

    * Unresponsive to medical therapy with anti-thymocyte globulin and/or cyclosporine
  * Inborn errors of metabolism, including, but not limited to the following:

    * Hurler's syndrome
    * Adrenoleukodystrophy
    * Maroteaux-Lamy syndrome
    * Globoid cell leukodystrophy
    * Metachromatic leukodystrophy
    * Fucosidosis
    * Mannosidosis
  * Fanconi anemia documented by increased chromosomal fragility assays and meeting 1 of the following criteria (stratum closed to accrual):

    * Severe pancytopenia

      * Absolute neutrophil count less than 500/mm^3
      * Platelet count less than 20,000/mm^3
      * Hemoglobin less than 8 g/dL
    * Morphologic evidence of MDS with clonal chromosomal abnormalities
    * Leukemia transformation
  * Other marrow failure syndromes, including any of the following (stratum closed to accrual):

    * Blackfan-Diamond syndrome that is unresponsive to medical therapy
    * Kostmann's congenital agranulocytosis unresponsive to medical therapy
    * Congenital amegakaryocytic thrombocytopenia
    * Thrombocytopenia absent radius
  * Combined immune deficiencies including, but not limited to the following:

    * Severe combined immunodeficiency (SCID)
    * Wiskott-Aldrich syndrome
    * Leukocyte adhesion defect
    * Chediak-Higashi disease
    * X-linked lymphoproliferative disease
    * Adenosine deaminase deficiency
    * Purine nucleoside phosphorylase deficiency
    * X-linked SCID
    * Common variable immune deficiency
    * Nezeloff's syndrome
    * Cartilage hair hypoplasia
    * Reticular dysgenesis
* No active CNS leukemia (cerebrospinal fluid with WBC greater than 5/mm^3 and malignant cells on cytospin)
* No SCID patients who do not require cytoreduction
* No dyskeratosis congenita
* No primary myelofibrosis
* No grade 3 or greater myelofibrosis
* Familial erythrophagocytic lymphohistiocytosis patients must not have any of the following:

  * Abnormal brain MRI
  * Neurologic symptoms
  * Lymphocytes and monocytes greater than 7/mm^3 in the cerebrospinal fluid
* No available 5/6 or 6/6 HLA-matched related donor

PATIENT CHARACTERISTICS:

Age

* 55 and under (over 18 closed to accrual)

Performance status

* Karnofsky 70-100% OR
* Lansky 50-100% (patients under 16 years old)

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* SGOT less than 5 times upper limit of normal
* Bilirubin less than 2.5 mg/dL

Renal

* Creatinine normal for age OR
* Creatinine clearance or glomerular filtration rate greater than 50% of lower limit of normal

Cardiovascular

* LVEF greater than 40% at rest and must improve with exercise* OR
* Shortening fraction greater than 26%* NOTE: *If symptomatic

Pulmonary

* DLCO greater than 45% of predicted* (corrected for hemoglobin)
* FEV_1 and FEC greater than 45% of predicted (corrected for hemoglobin) OR
* Room air oxygen saturation greater than 85%* NOTE: *If symptomatic

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled viral, bacterial, or fungal infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 12 months since prior allogeneic stem cell transplantation with cytoreductive preparative therapy
* More than 6 months since prior autologous stem cell transplantation

Chemotherapy

* See Biologic therapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior enrollment on this study
* No continuous life support (e.g., mechanical ventilation) within 1 year after study transplantation (for patients with inborn errors of metabolism)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-01; Primary Completion 2003-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Study Chair — Roswell Park Cancer Institute
Locations (25):
- United States (25):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Medical Center, University of California San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Children's Medical Center of Dallas, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington